CLINICAL TRIAL: NCT05515510
Title: Acceptance and Efficacy of a Digital Application in Promoting Evidence Based Oral Hygiene Knowledge Among Parents to Control Early Childhood Caries
Brief Title: Acceptance and Efficacy of a Digital Application Among Parents to Control Early Childhood Caries
Acronym: FU-APP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BB-097/20
Record Dates: First submitted 2021-05-05; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Early Childhood Caries; Oral Hygiene; Oral Health
Keywords: digital application; parental knowledge; parental behaviour; self-reported practices; self-reported attitude

STUDY DESIGN:
Intervention Model Description: Two arm, care-based, controlled, randomized clinical trial (RCT) using questionnaires and intraoral assessment.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Oral health prevention recommendations (frequency of brushing, technique, diet counselling, fluoride use, etc.) will be provided as usual by the dentist (verbal/oral) according to the current German "Ratgeber 2020" (KZBV,2029), which are implemented as standard oral health recommendation at the Department of Preventive and Pediatric Dentistry of Greifswald University.
  Parents in the control group will be ask after the intervention, and at the recalls (between 2 and 12 weeks and 3 months), to answer a questionnaire in order to determine their knowledge, behaviour, attitudes and related oral health practices.
  Interventions: Other: Oral health recommendations
- Test (Experimental): Oral health recommendations will be provided according to the current German "Ratgeber 2020" (KZBV,2029), which are implemented as standard at the Department of Preventive and Pediatric Dentistry of Greifswald University. Test arm receives this information with a digital application (FU-APP) in addition to the established oral health recommendation/instruction according to the current German "Ratgeber 2020" (KZBV,2020). After the intervention and at the recalls (between 2 and 12 weeks and 3 months), parents will be asked to answer two questionnaires in order to determine their FU-APP acceptance, knowledge, behaviour, attitudes and related practices.
  Interventions: Other: FU-APP; Other: Oral health recommendations

INTERVENTIONS:
Other: FU-APP — FU-APP is a web-based application using the guidelines and oral health recommendations provided by the current German "Ratgeber 2020". It provides information related to oral health care for the parents of children between 6 to 72 months of age. An account was made on a certified online web-development platform and an application was developed on it.
  This application serves as a practical guide for the parents of children under 6 years of age. It provides all the essential German guidelines related to first dental visits, expected dental findings, practical brushing technique steps, plaque disclosing activity, motivational brushing video, nutritional facts and behavioral habits to be avoided. It is a complete package of essential information and with high quality content that promotes prevention of ECC at an early age.
  Arms: Test
Other: Oral health recommendations — Oral health recommendations provided as usual (verbal/oral) according to the current German "Ratgeber 2020"

SUMMARY:
Few educational oral health applications, directed to the preschool children under the age of six years are available world-wide. The overall aim of this study is to evaluate the acceptance and efficacy of a digital application in improving evidence based oral hygiene knowledge among parents of young children to control Early Childhood Caries (ECC).

This study is split into two parts, the first one is aimed to understand the acceptance, usability and parental perception about a digital application being used to promote the evidence based oral hygiene knowledge among parents of young children to control ECC.

In a second phase (randomised clinical trial) the additional effect and acceptance of the digital application, and efficacy in improving parental knowledge, behaviour and self-reported practices/attitudes related to the oral health preventive measures will be presented.

DETAILED DESCRIPTION:
This two arm randomized cohort study is being undertaken at the Department of Preventive and Pediatric Dentistry at the University of Greifswald. Assessment of eligibility and application of intervention will be carried out by a single investigator (JH).

This study is being conducted in total in two phases. In the first, pilot phase - the digital application design, acceptance and parental perception will be assessed with the help of a questionnaire. In the second phase a two-arm controlled randomized clinical trial (RCT) will be conducted to assess the acceptance and efficacy of the application in improving parental knowledge, behaviour and self-reported practices/attitudes related to the oral health preventive measures. Clinically oral hygiene status and caries status of the participant children will be recorded too. The total appointment duration will also be measured.

Intervention:

Pilot study: After receiving the informed consent from the parents, the FU-APP digital application was shown to the parents attending the Department of Preventive and Pediatric Dentistry at the University of Greifswald for an oral health check-up on a tablet-PC. Once the parents have gained the experience of using the application and viewing the content, they were asked to fill out a user-acceptability questionnaire.

RCT: After receiving the informed consent from the parents, the child was seated on the dental chair for a normal check-up and the parents received the intervention according to the assigned arm in the form of information delivered. The information was based on the oral hygiene recommendations that followed the current German guidelines (counselling in diet, brushing instructions, and fluoride varnish application, nutrition and behavioural habits) according to the age of the child (Bundeszahnärztekammer 2020). Subsequently, parents in the test arm received additional information with the help of the web-based application (FU-APP) on a tablet-PC. Once the parents gained the experience of using the application and viewing the content, they were asked to fill out a knowledge-testing questionnaire in order to compare the knowledge at a follow up appointment. Parents in the control group also were asked to fill out the Questionnaire. Clinically oral hygiene status and caries status of the participant child were also recorded. For both arms, the follow-up visits took place 2 to 4 weeks and 3 months later and consisted of the same sequence of steps for the given intervention with modified questions included in the questionnaire to compare the improvement in oral health knowledge and the clinical records were recorded again to assess the improvement levels in the oral hygiene status.

Hypothesis:

The acceptance, usability and parental perception of a digital application (FU-APP) developed to promote evidence based oral hygiene knowledge among parents of young children to control ECC is positive and there is an additional positive effect in improving parental knowledge, behavior and self-reported practices/attitudes related to the oral health preventive measures while testing the efficacy of the FU-APP.

Application development:

An account is made on a certified online web-development platform and an application is developed on it. It will provide information related to oral health care for the parents of children between 6 to 72 months of age. FU application will be a web based application using guidelines and recommendations provided by the current German "Ratgeber 2020".

Sample size calculation:

Pilot study: Purposive sample including N = 20 parents of medically fit children aged between 6 months to 72 months.

RCT: The sample size was calculated assuming a difference of 0,5 between groups at follow-ups, setting α=5% and power (1-ß)=0.80 resulting in 28 children for every group. Adding an expected drop-out of 15%, a total sample size of 33 in every group (test and control) is needed.

Randomisation and allocation concealment:

Participants will be randomised through a computer-generated random-number list with allocation concealment to 1 of the 2 arms. Proper allocation concealment will be assured by a second investigator (RS), different to the investigator in charge of participants recruiting (JH). This investigator will have no possibility of knowing, which participant will go in which group avoiding influence on the randomisation.

Statistical analysis:

Part 1 - Pilot Data was primarily recorded on a spreadsheet Microsoft Excel (2017), then analysed using SPSS version 27. Spearman's correlation coefficient was applied to assess the strength of association between overall satisfaction and usage, acceptance, content and usefulness of the FU-App. Kruskal-Wallis analysis of variance and the non-parametric Mann-Whitney U test were applied to assess differences between FU category and overall satisfaction. P-value≤0.05 was taken as statistically significant.

Part 2 - Normality was checked for quantitative variables. Comparisons between the test and control were done using independent samples t-test, or Mann-Whitney U test for quantitative variables (according to the variable normality), while comparisons of qualitative variables were done using chi-square and Fisher exact tests, with Monte Carlo correction whenever indicated. Comparing the baseline and follow-up in each group was done using Wilcoxon signed rank and Mc-Nemar tests. Significance was inferred at p value <0.05. Data were analysed using IBM-SPSS for Windows (v. 23.0).

Quality assurance information:

Quality Assurance consisted of multiple steps in order to maintain a standard protocol during the study. As a first step, standard guidelines were set up for the data collection process through consensus by FU-Team. Secondly a detailed recruitment plan was developed to strategize and be aligned on the recruitment and data collection. Lastly the final step was to monitor and evaluate the process in the study field during the data collection and along with it identify the areas of improvement to strengthen the study further.

Standard procedures were used to ensure accurate and consistent measurements throughout the study. Standardized training was done in order to be familiar with the navigation of the FU-APP. Principal investigator (JH) was trained to conduct recruitment, measurement, and data collection for the RCT. The Principal investigator (JH) participated in a Quality Assurance (QA) training before starting the recruitment process. The training reviewed all data collection components and consisted of standardized measurements to minimize error. The training held before the follow-up sessions also included a mock data collection session.

The collected data information and documents were stored securely in the cabinets at the University Department. The consent forms and questionaries were filed properly in a customized folder designed and allocated to each recruited study participant. At the follow up appointment further documents were filed in the same individualized folder ensuring that each study participant had a customized protected folder and all quality assurance protocols are met. Only the principal investigator and study supervisors had the access to study participant's customized folders. Each study participant also received a copy of consent form and the confirmation form of willingness to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Parents can fully understand German language.
* Parents of medically fit children aged 6 months - 72 months.
* Parents/children who attend the Department of preventive and Pediatric Dentistry of the University of Greifswald for an oral health check-up.
* Willingness to participate in the study.

Exclusion Criteria:

* Parents who visit the Department of preventive and Pediatric Dentistry of the University of Greifswald for an emergency treatment or pain.
* Parents who decline to participate in the study.

Ages: 6 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Acceptance of the digital application | Baseline
  The pre-tested questionnaire will be used to test the overall acceptance level of the FU-APP. Answers will be as 5-point- Likert Scale (Completely agree, partially agree, neutral, partially disagree, completely disagree) presented.
  The questionnaire includes different categories: usage, acceptance, content description, usefulness and satisfaction.
Change in knowledge, behaviour and self-reported practices/attitude related to oral health preventive measures. | 2-4 weeks, and 3 months
  The questionnaire will be used to test change in knowledge, behavior and self-reported practices, attitude related to oral health preventive measures after having used the FU-APP. The options will be provided in the form of multiple choice.
Change in acceptance of a digital application | 2-4 weeks, and 3 months
  The questionnaire will be used to test the overall acceptance level (usage, content description, usefulness and satisfaction) of the FU-APP. Answers will be as 5-point- Likert Scale (Completely agree, partially agree, neutral, partially disagree, completely disagree) presented.

SECONDARY OUTCOMES:
O'Leary Plaque Index | Baseline and 3 months
  Visual assessment of plaque covered surfaces following application of a disclosing solution. The number of positively scored surfaces is divided by the total number of tooth surfaces evaluated, and the result is multiplied by 100 to express the index as a percentage.
Papilla Bleeding Index (PBI) | Baseline and 3 months
  To assess the severity of gingival inflammation in individual patients. Bleeding is provoked by sweeping the sulcus using a blunt periodontal probe under light finger pressure from the base of the papilla to its tip along the tooth's distal and mesial aspects. After 20-30 seconds, when a quadrant has been completely probed, the intensity of bleeding is scored in four grades and recorded on the chart.
  The sum of the recorded scores gives the "bleeding number." The PBI is calculated by dividing the bleeding number by the total number of papilla examined.
dmft caries index | Baseline and 3 months
  Caries experience for a child is expressed as the total number of teeth or surfaces that are decayed (d), missing (m), or filled (f). The dmft index expresses the number of affected teeth in the primary dentition, with scores ranging from 0 to 20 for children.

CONTACTS AND LOCATIONS:
Overall Officials: Jameela Abdul Haq, MSc, Principal Investigator — Universitätmedizin Greifswald
Locations (1):
- Universitätmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The German "Ratgeber 2020" (Bundeszahnärztekammer 2019) — https://www.kzv-sh.de/wp-content/uploads/2016/12/broschuere-fruehkindliche-karies-ecc.pdf